CLINICAL TRIAL: NCT03231618
Title: The Intervention Study of Dietary Intake on Energy Expenditure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Xu Lin, Principal Investigator, Chinese Academy of Sciences
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ChineseAS-201709
Record Dates: First submitted 2017-07-21; First posted 2017-07-27 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Healthy and Overweight/ Obesity Males
Keywords: dietary intake; cross-over intervention; energy expenditure
MeSH Terms: interventions — Diet, Fat-Restricted; Diet, Carbohydrate-Restricted

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal weight group (Experimental): 20 normal-weight males taking 3 types of assigned diets in random orders
  Interventions: Dietary Supplement: 1. Low-fat and high-carbohydrate diet; 2. High-fat and low-carbohydrate diet; 3. High-protein and low-fat diet
- Overweight/ obesity group (Experimental): 20 overweight/ obesity males taking 3 types of assigned diets in random orders
  Interventions: Dietary Supplement: 1. Low-fat and high-carbohydrate diet; 2. High-fat and low-carbohydrate diet; 3. High-protein and low-fat diet

INTERVENTIONS:
Dietary Supplement: 1. Low-fat and high-carbohydrate diet; 2. High-fat and low-carbohydrate diet; 3. High-protein and low-fat diet — Every participate was provided with 3 types of diets in random order

SUMMARY:
This study is a randomized crossover (2 × 3) dietary intervention. 40 male volunteers(20 normal weight, 20 overweight / obesity, no other serious disease or metabolic abnormalities) aged 18-45 years are required to take 3 kinds of isocaloric diets with different amounts of macronutrients: low-fat high-carbohydrate diets, low-carbohydrate high-fat diets and high-protein low-fat diets. The comparison is made within subject before and after the test meal. Each subject takes 6 meals of 3 kinds of diets on 6 separate days with a washout period between different diets. The study protocol was approved by the Ethics Committee of Shanghai Institutes for Biological Sciences and all participants provided written informed consents. The study is the first to investigate among overweight / obesity and normal weight in China to clarify:

1. the relationship between the proportion of macronutrients in diets and the energy metabolism efficiency.
2. the main genetic and non-genetic factors that impact individual energy metabolism, the characteristics of metabolic profiling and relative regulatory pathways.

DETAILED DESCRIPTION:
With the largest population of obesity and diabetes, China is suffering from heavy burden of obesity and major complications such as cardiovascular disease, type 2 diabetes and other major metabolic diseases ,which have become the major cause of disease death and continued to endanger the public health. In order to curb the incidence of obesity and its complications, more effective strategies are required to "prevent the move forward." With the arrival of "precise nutrition" era, precise weight management strategy for different sub-groups has become a hotspot of international research in this field.

Healthy diet and lifestyle are worldwide recognized as the most important and effective ways of preventing chronic metabolic diseases such as obesity. Recently, different combinations of macronutrients including "low-fat + high carbon", "low carbon + high fat", and "high protein + low fat" draw much more attention instead of restriction on the total energy intake in the study of diet weight reduction strategy. However, it is noteworthy that most studies are focused on groups and conducted on the Western population. Studies of different dietary structure, genetic background and metabolic phenotypes of energy metabolism are still scarce, and data of Chinese population are lacking in this field.

This study intends to provide 40 male volunteers aged 20-45 (20 normal weight, 20 overweight / obesity, no other serious illness or metabolic abnormalities) with three diets with different levels of macronutrients (low-fat + high-carbon foods, low-carbon + high-fat foods, and high-protein + low-fat foods) to 1) clarify the relationship between the ratio of macronutrients in diets and the energy metabolism efficiency; 2) investigate the effect of major genetic and non-genetic factors (age, obesity, adipose distribution and thyroid hormone) and metabolomics profiles on individual energy metabolism; 3) explore novel metabolic regulation networks. Ultimately, this study will provide basic data for discovering the energy metabolism efficiency of different dietary intervention and major genetic and non-genetic determinants, metabolic profile characteristics and regulatory pathways.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects, aged 18-45 years
* 20 normal weight (18.5≤ BMI<24) and 20 overweight / obesity (BMI ≥24)
* No participating in other clinical studies within previous 3 months

Exclusion Criteria:

* Alcoholic (100 grams of alcohol per drink, or 250 grams of rice wine, or 5 bottles of beer, ≥ 5 times a week)
* Diabetic patients or the use of insulin, hypoglycemic agents
* Taking antihypertensive drugs (diuretics, β blockers drugs, etc.) or lipid lowering drugs (class "bite", bile acids, statins, etc.) at present or once (within 6 months before the experiment)
* Having serious cardiovascular and cerebrovascular diseases at present or before, may interfere with the normal operation of the experiment (such as heart failure, myocardial infarction, cerebral infarction, acute myocarditis, severe arrhythmia, receiving interventional therapy, etc.)
* Having severe gastrointestinal diseases that affect food digestion and absorption, such as severe diarrhea in the past 3 months (3 or more times per day and lasting for 3 days or more); severe constipation in the past 3 months (2 times a week or less, accompanied by difficulties in defecation)
* Having received drug treatment over the past 3 months due to the following diseases: cholecystitis, gastrointestinal ulcers; urinary tract infection, acute pyelonephritis, cystitis; having undergone any surgery, in addition to appendicitis, hernia surgery; having taken or taking drugs that will affect the digestion and absorption system
* Attempting to change weight recently(weight loss, being on a diet, or weight gain)
* Subjects with severe liver and kidney disease (alanine aminotransferase, serum creatinine exceeded 1.5 times of the normal range set by the hospital)
* Subjects with severe thyroid disease (hyperthyroidism or hypothyroidism) or pituitary disease
* Subjects with anemia (hemoglobin <120 g per liter)
* Subjects with cancer or who have received radiotherapy or chemotherapy within five years
* Having any mental illness; epilepsy patients or receiving antiepileptic treatment; using antidepressants
* Suffering from AIDS, hepatitis A, hepatitis B or other infectious diseases
* Physical disability

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Respiratory Quotient | 1 hour after meal
  Respiratory quotient was measured in a metabolic chamber

SECONDARY OUTCOMES:
Heart Rate | 1 hour after meal
  Heart rate (bpm) was measured by automatic heart rate meter
Glucose | 2 hour after meal
  Blood glucose (mg/dl) was measured using a automatic biochemical analyzer
Triglyceride | 2 hour after meal
  Blood triglyceride (mg/dl) was measured using a automatic biochemical analyzer

CONTACTS AND LOCATIONS:
Overall Officials: Xu Lin, Principal Investigator — Institute for Nutritional Sciecnes, Chinese Acadamy of Sciences
Locations (1):
- Institute for Nutritional Sciences, Chinese Academy of Sciences, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sun L, Lin X. Reply to KR Short. J Nutr. 2022 Aug 9;152(8):2005-2006. doi: 10.1093/jn/nxac139. No abstract available. PMID 35849706
- [Derived] Xiong Q, Sun L, Luo Y, Yun H, Shen X, Yin H, Chen X, Lin X. Different Isocaloric Meals and Adiposity Modify Energy Expenditure and Clinical and Metabolomic Biomarkers During Resting and Exercise States in a Randomized Crossover Acute Trial of Normal-Weight and Overweight/Obese Men. J Nutr. 2022 Apr 1;152(4):1118-1129. doi: 10.1093/jn/nxac006. PMID 35020917